CLINICAL TRIAL: NCT07082751
Title: Prognostic Model for Metabolic Dysfunction-associated Steatotic Liver Disease Related Cirrhosis
Brief Title: Prognostic Model for MASLD Related Cirrhosis
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Vice president of hospital, Beijing Friendship Hospital
Other Study IDs: 2025-P2-166-01
Record Dates: First submitted 2025-06-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease; Compensated Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MASLD-related compensated cirrhosis: MASLD-related compensated cirrhosis confirmed by histopathology or clinical diagnosis
  Interventions: Behavioral: Lifestyle Guidance

INTERVENTIONS:
Behavioral: Lifestyle Guidance — Lifestyle Guidance

SUMMARY:
This study enrolled 228 patients with MASLD-related cirrhosis confirmed by histopathology or clinical diagnosis. Follow-up was conducted every 3-6 months. The primary endpoint was cumulative incidence of liver-related events (including decompensation events, hepatocellular carcinoma, liver transplantation, and liver-related mortality) and all-cause mortality. Secondary endpoints included cumulative incidence of metabolic events and changes in non-invasive fibrosis markers.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18 and 80 years (inclusive) who understand and sign informed consent forms; 2. Compensated MASLD-related cirrhosis diagnosis(meet one of the following conditions):

1. The liver biopsy during the screening period (liver biopsy within 6 months of screening is acceptable) showing cirrhosis with steatohepatitis according to the Non Alcoholic Fatty Liver Disease Clinical Research Network (NASH-CRN) scoring system, and there is no evidence of competitive aetiology.
2. The liver biopsy during the screening period (liver biopsy within 6 months of screening is acceptable) showing cirrhosis with steatosis (no steatohepatitis) according to NASH-CRN scoring system, and there is no evidence of competitive aetiology. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including overweight/obesity and/or prediabetes/type 2 diabetes mellitus (T2DM).
3. Historical biopsy showed steatohepatitis, and now diagnosed with cirrhosis through non-invasive tests or clinical criteria (see criterion (6)-1)). There is no evidence of competing aetiology. There is at least 1 coexisting or history of metabolic comorbidity.
4. Historical biopsy showed steatosis (no steatohepatitis), and now diagnosed with cirrhosis through non-invasive tests or clinical criteria (see criterion (6)-1)). There is no evidence of competing aetiology. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including overweight/obesity and/or prediabetes/type 2 diabetes mellitus (T2DM).
5. 'Cryptogenic cirrhosis' (with no evidence of hepatic steatosis on both histopathology and imaging). There is no evidence of competing aetiology. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including overweight/obesity and/or prediabetes/type 2 diabetes mellitus (T2DM).
6. MASLD-related cirrhosis is defined based on the following criterias:

   a. Cirrhosis is defined based on one of the following non-invasive tests(NITS): i: MRE ≥ 5kPa or VCTE-LSM ≥ 20kPa; ii:VCTE ≥15 kPa and <20 kPa and 1 of the following: MRE≥4.2kPa or Agile4≥0.565 or Platelets≤150,000/µL; iii: VCTE <15 kPa and 2 of the following: MRE≥4.2kPa or Agile4≥0.565 or Platelets≤150,000/µL; b. Current or previous imaging examinations have diagnosed fatty liver or controlled attenuation parameter (CAP)≥288dB/m or magnetic resonance imaging proton density fat fraction (MRI-PDFF)≥5%.

   c. There is no evidence of competing aetiology; d. There are at least 2 coexisting metabolic comorbidities or history of metabolic comorbidities, including overweight/obesity and/or prediabetes/type 2 diabetes mellitus (T2DM).

   Exclusion Criteria:
   * 1. Other chronic liver diseases (including but not limited to viral hepatitis, alcoholic liver disease, drug-induced liver injury, autoimmune liver disease, Wilson's disease, hemochromatosis, etc.) 2. There has been a continuous history of heavy drinking for 3 months or more current or rencent 5 years (heavy drinking is defined as >20 g/day in women and >30 g/day in men); Or researchers can not reliably quantify alcohol consumption.

     3. Hepatic decompensation events (including ascites, esophageal and gastric variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, spontaneous bacterial peritonitis, etc.) or hepatocellular carcinomaor.

     4. Previous (<5 years before screening) treatment for obesity with surgery; 5. Have obesity induced by other endocrinologic disorders (i.e. Cushing Syndrome) genetic diseases; 6. Secondary factors that can cause liver steatosis, such as malnutrition, medication, genetic metabolic diseases, etc.

     7. Positive for human immunodeficiency virus (HIV) infection; 8. History of drug use or abuse of drugs within the 12 months prior to screening.

     9. Pregnant or lactating women; 10. Researchers believe that patients who are not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MASLD related cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
composite endpoint | 5 years
  cumulative incidence of liver-related events (including decompensation events, hepatocellular carcinoma, liver transplantation, and liver-related mortality) and all-cause mortality.

SECONDARY OUTCOMES:
Metabolic Diseases | 5 years
  Number of participants with metabolic disease, including Type 2 Diabetes Mellitus (T2DM), Hypertension, Dyslipidemia
Cardiovascular Diseases (CVD) | 5 years
  Number of participants with CVD, including Coronary heart disease, Stroke, Heart failure, Atrial fibrillation
Non-Liver Tumors | 5 years
  Number of participants with non-liver tumors, including colorectal adenoma/adenocarcinoma, gastric cancer, esophageal cancer, pancreatic cancer, gallbladder cancer, lung cancer, prostate cancer, hematological malignancies and so on
non-invasive tests | 5 years
  changes in non-invasive test, including MRE, MRI-PDFF, LSM, CAP, APRI, FIB-4, NFS, Agile 4

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing University of Chinese Medicine Dongfang Hospital, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Capital Medical University, Beijing, China
  - Beijing Luhe Hospital, Capital Medical University, Beijing, China
  - Beijing Tsinghua Changgung Hospital, Beijing, China
  - Beijing Youan Hospital, Capital Medical University, Beijing, China
  - Peking University People's Hospital, Beijing, China
  - Tianjin Second People's Hospital, Tianjin, China
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, C

IPD SHARING:
Plan to Share IPD: Yes
Patient Demographics, Anthropometrics, Serological, and Imaging Data, and Liver Biopsy Scores
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the project finished
Access Criteria: ask the principle investigator